CLINICAL TRIAL: NCT03145948
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ABBV-553 in Healthy Volunteers and in Subjects With Psoriasis and Efficacy of ABBV-553 in Subjects With Psoriasis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ABBV-553 in Healthy Volunteers and in Subjects With Psoriasis and Efficacy of ABBV-553 in Subjects With Psoriasis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety reason
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: M16-058
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
Keywords: Tolerability; Psoriasis; Pharmacokinetics; Safety; Healthy Volunteers
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental): Participants, who are healthy volunteers, receiving ABBV-553 dose A or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo
- Arm B (Experimental): Participants, who are healthy volunteers, receiving ABBV-553 dose B or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo
- Arm C (Experimental): Participants, who are healthy volunteers, receiving ABBV-553 dose C or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo
- Arm D (Experimental): Participants, who are healthy volunteers, receiving ABBV-553 dose D or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo
- Arm E (Experimental): Participants with psoriasis receiving ABBV-553 dose B or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo
- Arm F (Experimental): Participants with psoriasis receiving ABBV-553 dose C or placebo
  Interventions: Drug: ABBV-553; Drug: Placebo

INTERVENTIONS:
Drug: ABBV-553 — It is administered orally.
Drug: Placebo — It is administered orally.

SUMMARY:
This is a study to assess the pharmacokinetics, safety and tolerability of multiple ascending oral doses of ABBV-553 in healthy volunteers and the pharmacokinetics, safety, tolerability and efficacy of multiple ascending oral doses of ABBV-553 in participants with psoriasis under non-fasting conditions.

ELIGIBILITY:
Inclusion Criteria: - Male or female and between 18 and 55 years of age, inclusive, for Substudy 1, OR between 18 and 75 years of age, inclusive, for Substudy 2.

* If female, participant must be of non-child bearing potential defined as either:

  a. Postmenopausal: Age > 55 years with no menses for 12 or more months without an alternative medical cause. Postmenopausal: Age <= 55 years with no menses for 12 or more months without an alternative medical cause AND a follicle stimulating hormone (FSH) level >= 40 IU/L (OR) b. Permanently surgical sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Non-postmenopausal females must have a negative urine pregnancy test result at Screening, and a negative serum pregnancy test result on Day -2 or Day -1.
* Male participants who are sexually active with women of child bearing potential (WOCBP), even if the male participant has undergone a successful vasectomy, must agree to use condoms from Day 1 through at least 30 days after the last dose of study drug, and male participant agrees not to donate sperm at least 30 days after the last dose of study drug.
* Body Mass Index (BMI) >= 18.0 to <= 29.9 kg/m2 after rounding to the tenths decimal for Substudy 1 OR BMI >= 18.0 to <= 34.9 kg/m2 after rounding to the tenths decimal for Substudy 2. BMI is calculated as weight measured in kilograms (kg) divided by the square of height measured in meters (m).
* In the opinion of the Investigator, that the participant is in a condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead Electrocardiogram (ECG).
* Must voluntarily sign and date each informed consent form, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures and be willing to comply with the requirements of this study protocol.

Additional criteria for Substudy 2:

* Has a clinical diagnosis of chronic plaque psoriasis (with a disease duration of at least 6 months).
* Has a Psoriasis Area and Severity Index (PASI) score ≥ 12.
* Has a Static Physician's Global Assessment (sPGA) score ≥ 3.
* Has a Body Surface Area (BSA) affected by Ps ≥ 10%. Exclusion Criteria: - Male participant who is considering fathering a child or donating sperm during the study or through 30 days after the last dose of study drug.
* History of clinically significant sensitivity to any drug.
* History of epilepsy, any clinically significant cardiac (including any family history of long-QT syndrome or unexplained sudden death), respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of gastric surgery (except pyloromyotomy for pyloric stenosis during infancy), vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
* Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the start of confinement (Day -2 or Day -1) or oral anti-infectives within 14 days prior to the start of confinement (Day -2 or Day -1)..
* Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements on a regular basis.
* Use of any medications, vitamins and/or herbal supplements within the 2-week period prior to study drug administration. For Substudy 2, medications used to treat chronic, stable medical conditions are allowed during screening and participation in the study unless the medication is specifically prohibited.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Substudy 1: Maximum observed plasma concentration (Cmax) of ABBV-553 | Day 1
  Maximum observed plasma concentration (Cmax) of ABBV-553
Substudy 2: Maximum observed plasma concentration (Cmax) of ABBV-553 | Day 1
  Maximum observed plasma concentration (Cmax) of ABBV-553
Substudy 1: Time to Cmax (peak time, Tmax) | Day 1
  Time to Cmax (peak time, Tmax)
Substudy 2: Time to Cmax (peak time, Tmax) | Day 1
  Time to Cmax (peak time, Tmax)
Substudy 1: Area under the concentration time curve (AUC) from time zero to 24 hours after dosing | Day 1
  Area under the concentration time curve (AUC) from time zero to 24 hours after dosing
Substudy 2: Area under the concentration time curve (AUC) from time zero to 24 hours after dosing | Day 1
  Area under the concentration time curve (AUC) from time zero to 24 hours after dosing
Substudy 1: Observed plasma concentration at the end of the dosing interval (Ctrough) | Day 7 and Day 14
  Observed plasma concentration at the end of the dosing interval (Ctrough)
Substudy 2: Observed plasma concentration at the end of the dosing interval (Ctrough) | Day 28
  Observed plasma concentration at the end of the dosing interval (Ctrough)
Substudy 1: Apparent clearance (CL/F) | Day 14
  Apparent clearance (CL/F)
Substudy 2: Apparent clearance (CL/F) | Day 28
  Apparent clearance (CL/F)
Substudy 1: Volume of distribution (Vβ/F) | Day 14
  Volume of distribution (Vβ/F)
Substudy 2: Volume of distribution (Vβ/F) | Day 28
  Volume of distribution (Vβ/F)
Substudy 1: Fraction excreted unchanged in urine (fe) | Day 14
  Fraction excreted unchanged in urine (fe)
Substudy 1: Apparent renal clearance (CLR) | Day 14
  Apparent renal clearance (CLR)

SECONDARY OUTCOMES:
Substudy 2: Psoriasis Area and Severity Index (PASI) | Day 28
  Percent improvement in PASI from Baseline
Substudy 2: Self-Assessment of Psoriasis Symptoms (SAPS) scores | Day 28
  Psoriasis subjects participating in Substudy 2 will complete the questionnaire at the designated clinic.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (4):
- United States (4):
  - Anaheim Clinical Trials LLC /ID# 164101, Anaheim, California
  - Providence Clinical Research /ID# 163867, Toluca, California
  - Progressive Medical Research /ID# 163868, Port Orange, Florida
  - Abbvie Clinical Pharmacology Research Unit /ID# 163866, Grayslake, Illinois